CLINICAL TRIAL: NCT04947735
Title: Control of Myopia Using Peripheral Diffusion Lenses: Efficacy and Safety Study Extension
Brief Title: CYPRESS Efficacy and Safety Study Extension
Acronym: CYPRESS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SightGlass Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPRO-1802-002
Record Dates: First submitted 2021-06-18; First posted 2021-07-01 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Juvenile Myopia; Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- CYPRESS Extension Test Arm (Experimental): Single vision, impact resistant spectacle lenses; CYPRESS Test Arm 1 and CYPRESS Test Arm 2 will move into CYPRESS Extension Test Arm
  Interventions: Device: Novel spectacle lens design
- CYPRESS Extension Control Arm (Placebo Comparator): Single vision, impact resistant spectacle lenses; CYPRESS Control Arm remains in control lenses as the CYPRESS Extension Control Arm
  Interventions: Device: Spectacle lenses

INTERVENTIONS:
Device: Novel spectacle lens design — Use of single vision, impact resistant spectacle lenses may reduce the rate of progression of juvenile myopia
  Arms: CYPRESS Extension Test Arm
Device: Spectacle lenses — Single vision, impact resistant spectacle lenses
  Arms: CYPRESS Extension Control Arm

SUMMARY:
This is an open-label, controlled, multisite, two-arm parallel group clinical trial of 36-month duration to evaluate the continued safety and efficacy of SightGlass Vision Diffusion Optics Technology (DOT) Spectacles in reducing the progression of juvenile myopia.

ELIGIBILITY:
Inclusion Criteria:

* Previously a successfully completed participant in the CYPRESS study (NCT03623074) and having not exited this study for more than 30 days;
* Agree to wear the assigned spectacles constantly except for sleeping, swimming, or other activities in which spectacle wear would be dangerous or otherwise not possible (minimum of 10 hours per day);
* Willingness to participate in the trial for up to 3 years without contact lens wear;
* The subject's parent(s) or legal guardian(s) must read, understand and sign the Statement of Informed Consent and receive a fully executed copy of the form.

Exclusion Criteria:

* Known allergy to proparacaine, tetracaine, or tropicamide.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Axial length | 72 months
  Test vs. control axial length change from baseline
Spherical equivalent refraction (SER) | 72 months
  Test vs. control spherical equivalent refraction (SER) change from baseline

SECONDARY OUTCOMES:
Axial length | 42 months
  Change from baseline
SER | 60 months
  Change from baseline

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - Golden Optometric Group, Whittier, California
  - Omega Vision Center, PA, Longwood, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - Haik Humble, West Monroe, Louisiana
  - Advanced Eyecare PC, Raytown, Missouri
  - SUNY School of Optometry, New York, New York
  - Sacco Eye Group, Vestal, New York
  - Dunes Eye Consultants, Dakota Dunes, South Dakota
  - Total Eye Care, Memphis, Tennessee
  - Dr. Bridgitte Shen Lee (PI), Houston, Texas
  - William J Bogus, OD, FAAO, Salt Lake City, Utah
- Centre for Ocular Research and Education, Waterloo, Ontario, Canada